CLINICAL TRIAL: NCT06904924
Title: Study of Determinants of the Nutritional Composition of Donor Human Milk
Brief Title: Determinants of the Nutritional Composition of Donor Human Milk
Status: Not yet recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Banco de Leite Humano do Norte (Unknown); Centro Hospitalar De São João, E.P.E. (Other); Faculdade de Medicina da Universidade do Porto - CINTESIS (Unknown); Faculdade de Ciências da Nutrição e Alimentação da Universidade do Porto (FCNAUP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BLHN/ Pediatric Nutrition
Record Dates: First submitted 2025-03-17; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Human Milk Nutrition
Keywords: Donor human milk; Human milk nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Donor's human milk (DHM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Human milk donor: Mothers who donate human milk to the BLHN of the Centro Hospitalar de São João.

SUMMARY:
Human milk is the most complete and correct way to feed a newborn, as it provides all the nutrients and bioactive factors essential for adequate growth and neurodevelopment. In special circumstances, such as prematurity or illness, breast milk is not always available, and donor human milk (DHM) is an option. Some studies have reported growth retardation in babies fed DHM, probably due to the less adequate nutritional composition. There are several factors that contribute to changes in its nutritional composition. Among the various factors, the following are worth highlighting: wide variety of donors with different characteristics (e.g. gestational age, lactation phase, diet); inconsistency of the collection method; impact of milk processing, i.e. the pasteurization process.

As the Human Milk Bank of North (BLHN - Banco de Leite Humano do Norte) is the first in the North region of Portugal, and there are few studies developed in this area in Portugal, the present project aims to study the influence of the following factors on the composition of the DHM:

* Pasteurization process;
* Dietary habits of donors;
* Body composition of donors.

DETAILED DESCRIPTION:
Study design and sampling: observational study with a cross-sectional and prospective design. The sample will consist of mothers who donate human milk to the BLHN of the Centro Hospitalar de São João.

Data collection: in order to meet the objectives of the research project, a questionnaire was drawn up for the participants, to be administered on paper, in an interview format, in the context of an outpatient consultation.

The questionnaire lasts around 20 minutes and consists of sociodemographic information (age, household composition, marital status, nationality, educational qualifications, profession); personal history (pathologies, number of pregnancies and births, date of last birth, gender, age, birth weight and length of the newborn, presence of gestational diabetes, hypertension in pregnancy, pre-eclampsia, term or pre-term birth, twin pregnancy); anthropometric data and body composition of the donor; food frequency questionnaire; physical activity; nutritional composition of the donated milk before and after processing (pasteurization).

ELIGIBILITY:
Inclusion Criteria:

* Human milk donors at BLHN
* Informed consent of the participant

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Human milk donors from BLHN
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Energy of donated human milk | At baseline before pasteurization; at baseline after pasteurization.
  Determination of the energy composition of the donated human milk (kcal/100mL).
Total protein levels of donated human milk | At baseline before pasteurization; at baseline after pasteurization.
  Determination of the total protein levels of the donated human milk (g/100mL).
True protein levels of donated human milk | At baseline before pasteurization; at baseline after pasteurization.
  Determination of true protein levels of the donated human milk (g/100mL).
Fat levels of donated human milk | At baseline before pasteurization; at baseline after pasteurization.
  Determination of fat levels of the donated human milk (g/100mL).
Carbohydrates levels of donated human milk | At baseline before pasteurization; at baseline after pasteurization.
  Determination of carbohydrates levels of donated human milk (g/100mL).
Body mass index of the donor | At baseline
  Height (m) and weight (kg) at the beginning and at the end of pregnancy of the donor to calculate pre-pregnancy body mass index (BMI) (kg/m^2) and the post-pregnancy BMI (kg/m^2).
Gestational weight gain of the donor | At baseline
  Gestational weight gain (kg) by the donor.
Waist circunference of the donor. | At baseline
  Waist circunference (cm) of the donor.
Hip circunference of the donor | At baseline
  Hip circunference (cm) of the donor.
Assessment of the donors' eating habits | At baseline
  The dietary habits of the previous year will be assessed using a semiquantitative food frequency questionnaire (FFQ) validated for the Portuguese adult population.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário São João (CHUSJ), Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided